CLINICAL TRIAL: NCT03263403
Title: A Randomized Observer-blinded Controlled Non-inferiority Trial to Evaluate the Immunogenicity of Locally Manufactured Meningococcal ACWY Vaccine 'Ingovax ACWY' in Bangladeshi Healthy Adults.
Brief Title: Non Inferiority Trial of Locally Manufactured Meningococcal ACWY Vaccine 'Ingovax ACWY' in Bangladesh.
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Collaborators: Incepta Vaccine Limited (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PR-17068
Record Dates: First submitted 2017-08-20; First posted 2017-08-28 (Actual); Last update posted 2018-03-22 (Actual); Status verified 2018-03

CONDITIONS: Meningococcal Vaccine
Keywords: Meningococcal Vaccine; Ingovax ACWY; adults; Bangladeshi; immunogenicity

STUDY DESIGN:
Intervention Model Description: Eligible participants will be assigned to receive the Ingovax ACWY Vaccine and Quadri Meningo Vaccine, in a 1:1 ratio across the target population according to the randomization schedule. 44 participants will receive locally produced Ingovax ACWY and 44 participants of comparator groups will receive Quadri Meningo which is produced by BiO-MeD Private Limited.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Since the test and comparator drugs used in this clinical study have different package of vial, a double blind design is not appropriate. Study investigators along with study staffs involved in safety evaluation and laboratory analysis will be blinded regarding the assigned treatment of the participant. The vaccine administration team will be unblinded to the treatment assignment list. The vaccine administrator team members will not be involved in the evaluation of vaccine safety and laboratory analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Group (Experimental): 44 participants will be randomly assigned to the test group for receiving the locally produced meningococcal vaccine "Ingovax ACWY" (Incepta).
  Interventions: Biological: Ingovax ACWY
- Comparator Group (Active Comparator): 44 participants will be randomly assigned to the comparator group for receiving 'Quadri Meningo' (BiO-MeD Private Limited).
  Interventions: Biological: Quadri Meningo

INTERVENTIONS:
Biological: Ingovax ACWY — The pharmaceutical company in Bangladesh is now currently marketing meningococcal vaccine of Yuxi Walvax Biotechnology Co. Ltd which is filled finish by Incepta Vaccines Ltd. This fill finish meningococcal vaccine is already registered and licensed in Bangladesh. However, at present, no locally produced meningococcal vaccine is available in Bangladesh. Once this clinical trial is completed, it will then proceed for registration and licensure in Bangladesh. Ingovax ACWY is a freeze-dried preparation of the group-specific polysaccharide antigens from Neisseria meningitidis Group A, Group C, Group Y and Group W135. When reconstituted, the vaccine is a clear, colorless sterile solution for subcutaneous use.
  Arms: Test Group
Biological: Quadri Meningo — Meningococcal polysaccharide vaccine Quadri Meningo vaccine manufactured by BiO-MeD Private Limited. Quadri Meningo [Meningococcal Polysaccharide Vaccine, Groups A, C, Y and W-135 Combined] is a freeze-dried preparation of the Group-specific polysaccharide antigens from Neisseria meningitidis, Group A, Group C, Group Y, and Group W-135. After reconstitution with diluent, the vaccine is a clear colourless liquid.
  Arms: Comparator Group

SUMMARY:
This study will be a randomized observer -blinded controlled non-inferiority study to evaluate and compare the immunogenicity of locally produced Ingovax ACWY with Quadri Meningo on a total of 88 healthy adult participants (18-45 years of age). 44 participants will receive locally produced Ingovax ACWY and 44 participants of comparator groups will receive Quadri Meningo which is produced by BiO-MeD Private Limited. Vaccination will be done in Day 0 following the screening and pre-immunization blood sample collection and post-immunization blood will be collected at Study Day 30. Follow- up by home visit will be carried out from Study day 1-6 and clinic follow-up is scheduled upto Study day 90. The hypothesis of this study is: locally produced subcutaneous Meningococcal vaccine Ingovax ACWY is non inferior and immunogenic among adults in Bangladesh as compared to Quadri Meningo.

DETAILED DESCRIPTION:
Protocol Title: A randomized observer-blinded controlled non-inferiority trial to evaluate the immunogenicity of locally manufactured Meningococcal ACWY vaccine 'Ingovax ACWY' in Bangladeshi healthy adults.

Background:

1. Burden:

   Meningococcal disease is an infectious disease caused by Neisseria meningitidis or meningococcus, which may present clinically as meningococcemia or meningitis, or presence of both features. Meningococcal meningitis causes inflammation of the membranes covering the brain and spinal cord. Meningococcal meningitis or meningococcemia is a life-threatening disease. It affects adults, adolescents and children as well. Every year more than 1.2 million people are affected by meningitis. It causes approximately 120,000 deaths globally each year. It can cause severe brain damage and is fatal in 50% of cases if untreated. According to a review article on meningococcal disease in Asia, results from four retrospective hospital-based studies conducted in Bangladesh showed that N. meningitidis present up to 35% of positive cultures in all ages, and up to 18% in children aged <2 years with bacterial meningitis. At the International Centre for Diarrhoeal Disease Research in Bangladesh, of 628 blood and CSF samples, N. meningitidis was detected in 24•8% (n=156), of which 97•7% were serogroup A and the rest 2.3% were serogroup B between 1999 and 2006. Of the 156 N. meningitidis isolates, 89 (57%) were from blood and 67 (43%) from CSF. Meningococcemia occurs without meningitis in 5% to 20% among the meningococcal infections. Globally the case-fatality ratio of meningococcemia is up to 40%.

   Despite of prompt diagnosis and the availability of appropriate treatments, the diseases is still a threat to the people. In spite of getting antibiotic in time, one in ten infected people die within 2 days of their first symptoms, one in four survivors is left with long-term disabilities such as loss of limb (s), deafness, nervous system problems, or brain damage. The disease can be transmitted as long as the symptoms persist or until 24 hours of effective treatment have been started. Carriers without symptoms can transmit the disease for about 6 months. Moreover, the disease can easily spread from person to person by respiratory droplets of sneezing or coughing or by sharing utensils.
2. Knowledge gap:

   Several different bacteria can cause meningitis. Neisseria meningitidis is the one with the potential to cause large epidemics. There are 12 Serogroups of N. meningitidis that have been identified, 6 of which (A, B, C, W, X and Y) can cause epidemics. But only a single dose of vaccine can prevent this deadly disease. Meningococcal Polysaccharide Vaccine of four serogroups A, C, W and Y that can protect from meningococcal meningitis and other associated diseases. It is a highly immunogenic and tolerable meningococcal vaccine to prevent meningococcal disease. World Health Organization recommends that countries with a moderate or high rate of disease or with frequent outbreaks should routinely vaccinate. Currently there is no locally manufactured Meningococcal vaccine available in Bangladesh. The results of this study will provide information regarding the immunogenicity of the locally manufactured meningococcal vaccine.
3. Relevance:

   The study of this locally manufactured Meningococcal Vaccine (Incepta) 'Ingovax ACWY' among adults will be able to give us information regarding the safety and immunogenicity of the vaccine. To get registration of this own bulk and finished product, Incepta intends to conduct clinical trials in human. Incepta has already conducted two Pre-clinical Studies at Reliance clinical research" in Mumbai, India. Toxicological evaluation of Meningococcal ACWY Vaccine (Ingovax) was conducted in Swiss albino mice and Sprague Dawley rats. No mortality or morbidity was observed in any of the animals in the control or the treated groups. No treatment related abnormal changes were observed in Clinical Signs, Body Weight, Food Consumption and Ophthalmological Examination. In the light of the above findings, No Observed Adverse Effect level (NOAEL) of Meningococcal ACWY Vaccine (Ingovax) is 50µg per rat or mouse. So, after successful completion of Preclinical study, the non-inferiority trail with this vaccine needs to be carried out with innovator product and move forward to licensure in Bangladesh. Currently there is no locally manufactured Meningococcal vaccine available in Bangladesh. Once this clinical trial is complete, it will then proceed for registration and licensure in Bangladesh. Thus the vaccine cost could be significantly reduced and save a large amount of foreign currency of Bangladesh Government.

   Hypothesis (if any): Locally produced subcutaneous Meningococcal vaccine Ingovax ACWY is non inferior and immunogenic among adults in Bangladesh as compared to Menomune® - A/C/Y/W-135.

   Objectives: The objective of this study is to

   Primary Objective:

   1.To evaluate and compare the immunogenicity of Ingovax ACWY' with Quadri Meningo in healthy adults in Bangladesh.

   Secondary Objective:

   1. To evaluate and compare the safety of locally produced Ingovax ACWY with Quadri Meningo.

   Methods:

   This will be a randomized observer -blinded controlled non-inferiority study on a total of 88 healthy adult participants (18-45 years of age). 44 Ingovax ACWY'0.5 ml (Test group) and 44 Quadri Meningo 0.5 ml (Comparator Group).

   Outcome measures/variables: To evaluate and compare the immunogenicity and safety of locally produced Ingovax ACWY' with Quadri Meningo vaccine.

   Primary end points:

   1. Assessment of proportion of participants showing seroconversion (defined as a ≥4-fold rise in SBA titers) vaccinated with either Ingovax ACWY Vaccine (Incepta) or Quadri Meningo vaccine (BiO-MeD Private Limited). The non-inferiority margin will be 10%.

   Secondary end points:
   1. To compare the GMTs between vaccines, and GMT ratios.
   2. Number of immediate reactions reported within 30 minutes after vaccination
   3. Number of solicited adverse events (prelisted in the participant's memory aid) occurring up to 7 days following vaccination.
   4. Number of unsolicited AEs up to 28days after vaccination.
   5. Occurrence of serious adverse events (SAEs) throughout the trial

ELIGIBILITY:
Inclusion Criteria:

1. Apparently healthy adult of 18 to 45 years of age.
2. Sex: Male, Female and Transgender
3. Apparently healthy based on a medical history taken prior to vaccination. Any underlying chronic illness must be documented to be in stable condition.
4. Women with child bearing potential must be non pregnant which will be confirmed by negative urine pregnancy test during screening and prior to vaccination on day 0 as well. Moreover, medical history will be taken thoroughly by study physician from the woman of childbearing age to completely exclude the probability of pregnancy.Women who are married and living with a partner must agree to use a reliable contraceptive method to prevent pregnancy until final follow-up following vaccination. However abstinence is also acceptable.

Exclusion Criteria:

1. Prior history of Meningitis infection or vaccination with any Meningococcal vaccine.
2. Prior history of taking any other polysaccharide vaccine (Pneumococcal Vaccine, Typhoid Vaccine) in last 6 months.
3. Receipt of investigational drugs or other investigational vaccines within 3 months prior to first injection with the study vaccine.
4. Recent febrile illness (within last two weeks).
5. Clinically significant abnormalities in screening hematology or serum chemistry, as determined by the Study Physician.
6. Known or suspected hypersensitivity to any component of Meningococcal ACWY polysaccharide vaccine.
7. Known or suspected impairment of immunologic function or recent use of immunomodulatory medications (e.g, systemic corticosteroids). Does not include topical and inhaled steroids.
8. Pregnant women, nursing mothers, and women planning to become pregnant within the study period.
9. Any condition which, in the opinion of the investigator, might interfere with the evaluation of the study objectives.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 88 (Actual)
Dates: Start 2017-08-21 (Actual); Primary Completion 2018-03-19 (Actual); Study Completion 2018-03-19 (Actual)

PRIMARY OUTCOMES:
Assessment of proportion of participants showing seroconversion (defined as a ≥4-fold rise in SBA titers) vaccinated with either Ingovax ACWY Vaccine (Incepta) or Menomune ® -A/C/Y/W-135 vaccine (Sanofi Pasteur Inc.). The non-inferiority margin will be | 30 days after administration of vaccine
  The test vaccine will induce similar seroconversion rates in compare to reference vaccine (defined as a ≥4-fold rise in SBA titers). This will be done by calculating the responder rate through comparing the pre and 30(±2) days post-vaccination serum bactericidal titres among Ingovax ACWY' or Menomune® - A/C/Y/W-135 vaccinated participants. The non-inferiority margin will be 10%. Serum bactericidal assay(SBA) titres and fold-rises will be logarithmically transformed prior to statistical analyses in order to better approximate normality.

SECONDARY OUTCOMES:
To compare the GMTs between vaccines, and GMT ratios. | 30 days after administration of vaccine
  Comparison of the geometric mean titre among the test and comparator group.
Number of immediate reactions reported within 30 minutes after vaccination | 30 minutes post vaccination
  After administration of study agents, participants will be requested to wait for at least 30 minutes at the vaccination sites to monitor for any solicited adverse events following vaccination.
Number of solicited adverse events (prelisted in the participant's memory aid) occurring up to 6 days following vaccination. | Post vaccination Day 1 to Day 6
  Participants will be monitored specifically for local adverse reactions (redness, swelling, pain, tenderness, induration and ecchymosis) and systemic reactions (headache, seizure, rash, arthalgia, myalgia, fever, nausea, vomiting, diarrhea, shivering, fatigue and malaise). These adverse events will be monitored actively for the first 6 days in all participants following vaccination.
Number of unsolicited AEs up to 28days after vaccination. | 28 days following vaccination
  Adverse events will be monitored passively up to 28 days post dose of IP administration.
Occurrence of serious adverse events (SAEs) throughout the trial | upto 90 days post vaccination
  serious adverse events that occurs from the beginning of the study up to the end (90 days after vaccination) will be reported using the Serious Adverse Event forms.

CONTACTS AND LOCATIONS:
Overall Officials: Firdausi Qadri, PhD, Study Director — International Centre for Diarrhoeal Disease Research, Bangladesh
Locations (1):
- Mohiul Islam Chowdhury, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hart CA, Thomson AP. Meningococcal disease and its management in children. BMJ. 2006 Sep 30;333(7570):685-90. doi: 10.1136/bmj.38968.683958.AE. No abstract available. PMID 17008668
- [Background] Hossain MA, Ahmed D, Ahmed T, Islam N, Breiman RF. Increasing isolations of Neisseria meningitides serogroup A from blood and cerebrospinal fluid in Dhaka, Bangladesh, 1999-2006. Am J Trop Med Hyg. 2009 Apr;80(4):615-8. PMID 19346387
- [Background] Vyse A, Wolter JM, Chen J, Ng T, Soriano-Gabarro M. Meningococcal disease in Asia: an under-recognized public health burden. Epidemiol Infect. 2011 Jul;139(7):967-85. doi: 10.1017/S0950268811000574. Epub 2011 Apr 15. PMID 21492496
- [Background] Crum-Cianflone N, Sullivan E. Meningococcal Vaccinations. Infect Dis Ther. 2016 Jun;5(2):89-112. doi: 10.1007/s40121-016-0107-0. Epub 2016 Apr 16. PMID 27086142
- [Background] Stephens DS, Greenwood B, Brandtzaeg P. Epidemic meningitis, meningococcaemia, and Neisseria meningitidis. Lancet. 2007 Jun 30;369(9580):2196-2210. doi: 10.1016/S0140-6736(07)61016-2. PMID 17604802
- [Background] Memish ZA. Meningococcal disease and travel. Clin Infect Dis. 2002 Jan 1;34(1):84-90. doi: 10.1086/323403. Epub 2001 Nov 20. PMID 11731951
- [Background] Control and prevention of meningococcal disease: recommendations of the Advisory Committee on Immunization Practices (ACIP). MMWR Recomm Rep. 1997 Feb 14;46(RR-5):1-10. PMID 9048846
- [Derived] Ahmed T, Tauheed I, Hoque S, Sarower Bhuyan G, Biswas R, Tarikul Islam M, Islam S, Amir Hossain M, Ahmmed F, Muktadir A, Muktadir H, Ahmed F, Karim M, Panday AS, Kundu Tanu T, Muktadir Rahman Ashik M, Rahad Hossain M, Shariful Bari S, Ahmed R, Masudur Rahman Mia M, Islam S, Khan I, Mainul Ahasan M, Chowdhury F, Rahman Bhuiyan T, Islam Chowdhury M, Qadri F. A phase 3 non-inferiority trial of locally manufactured Meningococcal ACWY vaccine 'Ingovax ACWY' among Bangladeshi adults. Vaccine. 2024 Oct 3;42(23):126063. doi: 10.1016/j.vaccine.2024.06.030. Epub 2024 Jun 18. PMID 38897895